CLINICAL TRIAL: NCT03829527
Title: Evaluation of the Treatment Approach ROBIN (Standardized Manual and Smartphone App) for Adolescents With High Risk for Developing a Psychotic Disorder
Brief Title: Evaluation of the Treatment Approach ROBIN
Acronym: Robin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: ETRo2017-00012
Record Dates: First submitted 2019-01-24; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Clinical High Risk for Psychosis
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychotherapy (Experimental)
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Psychological intervention combining a standardized treatment manual with a smartphone application

SUMMARY:
The prevention of schizophrenia and other psychotic disorders has led researchers to focus on early identification of individuals at Clinical High Risk (CHR) for psychosis and to treat the at-risk symptoms in the pre-psychotic period. Although at-risk symptoms such as attenuated hallucinations or delusions are common in adolescents and associated with a marked reduction in global functioning, the evidence base of effective interventions for adolescents at CHR state and even ﬁrst-episode psychosis is limited. To fill this gap, the clinicians from the early intervention center in Zurich have developed the treatment approach "Robin" (standardized manual and smartphone App) for adolescents with high risk for developing a psychotic disorder. The treatment approach is based on existing therapy strategies for adolescents with first episode of psychosis and the available recommendations for adults with at-risk symptoms. The evaluation aims firstly to compare the efficacy of "Robin" in 30 CHR adolescents aged 14-18 to an active control group (treatment as usual) from a previous study. Primary outcome measures will be at-risk symptomatology, comorbid diagnosis, functioning, self-efficacy and quality of life. For the prospective intervention condition (16 weekly individual sessions + a minimum 4 family sessions), help-seeking adolescents with CHR for psychosis, aged 14-18, will be recruited over three years. At-risk and comorbid symptoms, functioning, self-efficacy and quality of life are monitored at six time points (baseline, during the treatment period, immediately after intervention, and 6, 12, and 24 months later) and compared to the respective measures of the active control group.

ELIGIBILITY:
Inclusion Criteria:

* 1) At least two self-experienced and self-reported cognitive basic symptoms as assessed by the children-youth version of the Schizophrenia Proneness Interview Child and Youth Version (SPI-CY)
* and/or 2) at least one attenuated psychotic symptom for psychosis assessed by the Structured Interview for Prodromal Syndromes (SIPS)

Exclusion Criteria:

* a diagnosis of a psychotic disorder
* current substance or alcohol dependence
* insufficient German or English language ability
* low intellectual abilities with IQ <75

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in at risk symptoms over the different time points | Baseline (0 months); during the treatment (2 months), post-treatment (4 months), follow ups (6, 12, 24 months)
  According to a structured clinical interviews about the clinical high risk state(SIPS, SPI-CY)
Changes in comorbid symptoms over the different time points | Baseline (0 months); during the treatment (2 months), post-treatment (4 months), follow ups (6, 12, 24 months)
  According to a structured clinical interviews about the comorbid symptoms (M.I.N.I. Kid)
Changes in overall global functioning over the different time points | Baseline (0 months); during the treatment (2 months), post-treatment (4 months), follow ups (6, 12, 24 months)
  Measured by Global Assessment of Functioning Scale GAF. The Global Assessment of Functioning (GAF) is a numeric scale used by mental health clinicians and physicians to rate subjectively the social, occupational, and psychological functioning of an individual, e.g., how well one is meeting various problems-in-living. Scores range from 100 (extremely high functioning) to 1 (severely impaired).
Changes in the social and occupational functioning over the different time points | Baseline (0 months); during the treatment (2 months), post-treatment (4 months), follow ups (6, 12, 24 months)
  Measured by the Social and Occupational Functioning Assessment Scale SOFA . The SOFAS is a new scale that differs from the Global Assessment of Functioning (GAF) Scale in that it focuses exclusively on the individual's level of social and occupational functioning and is not directly influenced by the overall severity of the individual's psychological symptoms. The SOFAS is a global rating of current functioning ranging from 0 to 100, with lower scores representing lower functioning.
Changes in social functioning over the different time points | Baseline (0 months); during the treatment (2 months), post-treatment (4 months), follow ups (6, 12, 24 months)
  Measured by theGlobal Functioning: Social (GF: Social) scale The GF: Social scale assesses quantity and quality of peer relationships, level of peer conflict, age-appropriate intimate relationships, and involvement with family members. Emphasis is placed on age-appropriate social contacts and interactions outside of the family, with a particular focus on social withdrawal and isolation. The scales range from 1 till 10 (10 is the highest rating).
Changes in the quality of life over the different time points: MANSA | Baseline (0 months); during the treatment (2 months), post-treatment (4 months), follow ups (6, 12, 24 months)
  Self reported level of life quality measured with the Manchester Short Assessment of Quality of Life (MANSA). 16 questions are to be asked every time the instrument is applied. Four of these questions are termed objective and to be answered with yes or no. Twelve questions are strictly subjective. The satisfaction is rated on 7-point rating scales ( = negative extreme, 7 = positive extreme). The twelve items are in the end combined (summed) to get a total score about the life quality.
Changes in the self efficacy over the different time points: General Self-efficacy Scale (SWE) | Baseline (0 months); during the treatment (2 months), post-treatment (4 months), follow ups (6, 12, 24 months)
  Self reported level of self efficacy measured with the General Self-efficacy Scale (SWE). The General Self-Efficacy Scale is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life. The total score can vary between 10 (very low self-efficacy) and 40 (very high self-efficacy).

SECONDARY OUTCOMES:
Satisfaction with the treatment: questionnaire | 4 months (post-treatment)
  Subjective satisfaction with the therapy measured by a german questionnaire about the treatment satisfaction. The questionnaire is called "Fragebogens zur Beurteilung der Behandlung". Translation ins english is: Questionnaire about the treatment satisfaction.
  It contains 20 different questions about the treatment satisfaction on a rating scale from 0 till 5. So, the total score is between 0 (no treatment satisfaction) and 100 (highest treatment satisfaction).
7.Satisfaction with the smartphone application Robin Z: feedback form. | 4 months (post-treatment)
  Subjective satisfaction with the smartphone application measured by questionnaire regarding usability and subjective satisfaction with the app. The questionnaire was created by the study team, no standardized measurement tool is used. The questionnaire is a feedback form, that gives the study team qualitative information about the usability and satisfaction with the smartphone application. The only quantitive information that is gained from this questionnaire is the overall satisfaction with the application. The subjects can give a rating from 1 (lowest satisfaction) till 6 (highest satisfaction).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Department of Child and Adolescent Psychiatry and Psychotherapy, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fux L, Walger P, Schimmelmann BG, Schultze-Lutter F. The Schizophrenia Proneness Instrument, Child and Youth version (SPI-CY): practicability and discriminative validity. Schizophr Res. 2013 May;146(1-3):69-78. doi: 10.1016/j.schres.2013.02.014. Epub 2013 Mar 6. PMID 23473813
- [Background] Miller TJ, McGlashan TH, Rosen JL, Cadenhead K, Cannon T, Ventura J, McFarlane W, Perkins DO, Pearlson GD, Woods SW. Prodromal assessment with the structured interview for prodromal syndromes and the scale of prodromal symptoms: predictive validity, interrater reliability, and training to reliability. Schizophr Bull. 2003;29(4):703-15. doi: 10.1093/oxfordjournals.schbul.a007040. PMID 14989408
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Hall RC. Global assessment of functioning. A modified scale. Psychosomatics. 1995 May-Jun;36(3):267-75. doi: 10.1016/S0033-3182(95)71666-8. PMID 7638314
- [Background] Cornblatt BA, Auther AM, Niendam T, Smith CW, Zinberg J, Bearden CE, Cannon TD. Preliminary findings for two new measures of social and role functioning in the prodromal phase of schizophrenia. Schizophr Bull. 2007 May;33(3):688-702. doi: 10.1093/schbul/sbm029. Epub 2007 Apr 17. PMID 17440198
- [Background] Morosini PL, Magliano L, Brambilla L, Ugolini S, Pioli R. Development, reliability and acceptability of a new version of the DSM-IV Social and Occupational Functioning Assessment Scale (SOFAS) to assess routine social functioning. Acta Psychiatr Scand. 2000 Apr;101(4):323-9. PMID 10782554
- [Background] Priebe S, Huxley P, Knight S, Evans S. Application and results of the Manchester Short Assessment of Quality of Life (MANSA). Int J Soc Psychiatry. 1999 Spring;45(1):7-12. doi: 10.1177/002076409904500102. PMID 10443245
- [Background] Schwarzer, R., & Jerusalem, M. (1995). General Self-efficacy Scale. Measures in Health Psychology: A User's Portfolio. Causal and Control Beliefs, (2008), 35-37.
- [Derived] Traber-Walker N, Gerstenberg M, Metzler S, Joris MR, Karr M, Studer N, Zulauf Logoz M, Roth A, Rossler W, Walitza S, Franscini M. Evaluation of the Combined Treatment Approach "Robin" (Standardized Manual and Smartphone App) for Adolescents at Clinical High Risk for Psychosis. Front Psychiatry. 2019 Jun 6;10:384. doi: 10.3389/fpsyt.2019.00384. eCollection 2019. PMID 31244692